CLINICAL TRIAL: NCT04260048
Title: Impact of Hypothalamic Gliosis on Appetite Regulation and Obesity Risk in Children
Status: Completed | Type: Observational
Sponsor: University of Washington (Other)
Collaborators: Johns Hopkins University (Other); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Ellen Schur, MD, MS, Associate Professor, School of Medicine, University of Washington
Other Study IDs: SITE00000078; 1R01DK117623-01A1 (NIH)
Record Dates: First submitted 2020-01-28; First posted 2020-02-07 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Obesity, Childhood
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Permission to obtain and store a sample of whole blood to look at DNA in the future will be made.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Normal weight: Group defined based on BMI percentile for age and sex.
- Overweight: Group defined based on BMI percentile for age and sex.
- With obesity: Group defined based on BMI percentile for age and sex.

SUMMARY:
BEAM is a multi-site longitudinal cohort study of hypothalamic gliosis, central regulation of appetite and weight gain in children. Participants will be recruited from the community in the greater Seattle and greater Baltimore area. All participants will consent to enroll in the 24-month study during which they will complete 5 in-person study visits.

DETAILED DESCRIPTION:
The proposed 2-site research study uses a longitudinal cohort design in 102 children aged 9-11 yr. It will include for all participants baseline MRI and functional MRI, in-depth eating behavior testing, and measurement of hormone profiles. Serial measurement of weight and self-reported eating habits will occur over 2 yr, with a repeated MRI at 2 yr. The study aims to: 1) test if MBH gliosis is associated with impaired intake regulation and poor weight outcomes over 2 yr in children, 2) determine if CNS appetitive processing is negatively affected when evidence of MBH gliosis is present, and 3) test for other brain regions in which gliosis is present in association with excess adiposity in children. An exploratory aim will assess changes in gliosis in children over 2 yr and their relation to changes in body weight and adiposity.

ELIGIBILITY:
Inclusion Criteria:

* 9-11 y (at time of enrollment)
* BMI ≥ 15th percentile for age and sex

Exclusion Criteria:

* Significant Health conditions (e.g., type 2 diabetes)
* Documented cognitive disorder
* History of major weight loss of 10lbs or more, not due to illness, over the past year
* Eating disorder (e.g. anorexia, bulimia)
* Current use of medications known to alter appetite, body weight or brain response including: Anti-epileptics; Glucocorticoids; Antipsychotics; Stimulants for ADHD
* MRI contraindication (e.g. implanted metal, claustrophobia, inability to fit in MRI scanner)
* Weight >330 pounds (MRI limit)
* Severe food allergies, vegetarian, or vegan, or unable to eat study foods
* Currently in formal weight loss program

Ages: 9 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: A total of 102 participants (51 per site), age 9-11 years, will be recruited into 1 of three groups: Lean, Overweight, or Obese based on BMI percentile for age and sex.
Sampling Method: Non-Probability Sample
Enrollment: 101 (Actual)
Dates: Start 2020-02-21 (Actual); Primary Completion 2024-03-28 (Actual); Study Completion 2024-05-30 (Actual)

PRIMARY OUTCOMES:
Hypothalamic gliosis | 2 years
  Evidence of hypothalamic gliosis as measured by T2 relaxation time using MRI
Habitual dietary intake | 2 years
  Dietary intake in children by 24-hour dietary recalls
Obesity | 2 years
  Child BMI z-score calculated by the measures of height and weight

CONTACTS AND LOCATIONS:
Overall Officials: Ellen A Schur, MD, MS, Principal Investigator — University of Washington
Locations (2):
- United States (2):
  - Johns Hopkins University, Baltimore, Maryland
  - University of Washington, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No